CLINICAL TRIAL: NCT04541849
Title: Predicting Clinical Outcomes of Critically Ill Patients in Intensive Care Units With De-identification Database
Brief Title: Database for Predicting Clinical Outcomes of Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202004016RINB
Record Dates: First submitted 2020-08-30; First posted 2020-09-09 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients
  Interventions: Other: Critical Care

INTERVENTIONS:
Other: Critical Care — Critical care in the intensive care units

SUMMARY:
Australian and New Zealand Intensive Care Society (ANZICS) has built a Center of Outcome and Resource Evaluation (CORE) adult patients database (APD) of adult critically ill patients. ANZICS CORE APD has built an international collaboration of ICU database. National Taiwan University Hospital has joined this international collaboration and built the data according to the APD data dictionary with same value domain attributes and data element attributes. We retrospectively collected the data of patients discharged from the March 1, 2019 to June 30, 2022. Data of this database are permitted to study clinical problems and predict the clinical outcomes of these critically ill patients using statistical methods and machine learning techniques.

DETAILED DESCRIPTION:
Data of this database are permitted to study the following clinical issues: including delirium, sepsis, acute kidney injury, acute respiratory distress syndrome, disseminated intravascular coagulation, multiple organ injuries, nutrition, survival status, number of days on ventilators, need for renal replacement therapy, length of stays in intensive care unit, length of stay in hospital, and other relevant clinical outcomes. It is also planned to analyze the clinical prognosis of special disease subgroups and establish a prediction model according to the type of patient's disease.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients admitted to intensive care units

Exclusion Criteria:

* patients aged less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  mortality status at 30 days after admission to intensive care unit

SECONDARY OUTCOMES:
Length of stay in intensive care unit | Time of discharge from intensive care unit, a median of 2-7 days
  number of days in intensive care unite
Delirium | 48 hours
  Events of delirium within 48 hours after ICU admission
Acute kidney Injury | 48 hours
  Events of acute kidney injury within 48 hours
  Time Frame:
Length of stay in intensive care unit | Time of discharge from hospital, more than 1 day
  Number of days in intensive care unite
Disseminated intravascular coagulation | 48 hours
  Events of disseminated intravascular coagulation within 48 hours after ICU admission
Acute respiratory distress syndrome | 48 hours
  Events of acute respiratory distress syndrome within 48 hours after ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available according to the regulation of research ethic committee of National Taiwan University Hospital.